CLINICAL TRIAL: NCT05232942
Title: Monoclonal Antibody Duration of REsponse in MIgraine After Treatment Interruption: A Prospective National Study
Brief Title: Monoclonal Antibody Duration of REsponse in MIgraine After Treatment Interruption
Acronym: MADRE-MIA
Status: Recruiting | Type: Observational
Sponsor: Hospital Clínico Universitario de Valladolid (Other)
Responsible Party: Principal Investigator, David García Azorín, Headache Unit, Department of Neurology, Principal Investigator, Hospital Clínico Universitario de Valladolid
Other Study IDs: PI 20-1687
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Migraine; Headache, Migraine
Keywords: Treatment outcome; Evidence-based practice; Headache disorders, primary; Migraine; Treatment; Preventive treatment
MeSH Terms: conditions — Migraine Disorders; Headache Disorders, Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Studied group: The study population will consist of patients with diagnosis of episodic or chronic migraine who, under the criteria of their neurologist and according to the clinical practice guidelines and standard of care, receive treatment with monoclonal antibodies against CGRP (galcanezumab, fremanezumab or eptinezumab) or else its receptor (erenumab), with positive response, and discontinue the treatment.
  Interventions: Other: Headache calendar completion

INTERVENTIONS:
Other: Headache calendar completion — The patient will complete an in-paper or electronic calendar, depicting the presence/absence of headache, the median intensity and the need of acute medication.

SUMMARY:
Observational analytic study with a prospective cohort design. Patients with episodic and chronic migraine that have responded to monoclonal antibodies (mAbs) versus calcitonin gene-related peptide (CGRP) or its receptor with positive response will be included. A headache diary will be completed in a daily basis. The primary outcome will be the time elapsed between the discontinuation of the monoclonal antibody and the return to the clinical situation at the moment of the mAbs onset. The potential variables that may be associated with a more sustained benefit will be explored.

DETAILED DESCRIPTION:
Introduction:

The development of new preventive treatments represents a new era in the treatment of migraine. Different drugs have shown a reduction in the number of headache days, average intensity of pain and the need for symptomatic treatment in randomized, placebo-controlled trials; nonetheless, there are unanswered questions from clinical trials which are of a particular interest to routine clinical practice.

The duration of preventive treatments is not fully established, in the different clinical trials the duration of treatment ranged between 3, 6 or 12 months 3-12 . Additionally, it is known that the benefit of a preventive drugs may persist once interrupted, while in other cases, patients may return to the previous situation in a relatively short period of time. In the case of other preventive treatments, the therapeutic effect seems to be maintained for a longer period after the discontinuation of the treatment.

Preventive drugs targeting the Calcitonin gene-related peptide (CGRP) or its receptor have been approved. In Spain three of them (erenumab, galcanezumab and fremanezumab) are subsidized for the treatment of episodic migraine or chronic migraine in patients with at least 8 days of migraine per month and who have previously failed at least 3 preventive treatments. Still, the long-term duration of therapeutic effect once these treatments are suspended has not been clarified yet.

As the duration of the effect after discontinuing treatment and the optimal duration of treatment are not fully known, the present study aims to evaluate patients with migraine who have been treated with monoclonal antibodies. Additionally, the needed time to return to the situation prior to this treatment will be studied. The factors that may be associated with the duration of the benefit after the treatment discontinuation will be explored by using survival analysis methods.

Material and methods Observational study with a prospective cohort design. Patients with diagnosis of episodic or chronic migraine who, under the criteria of their neurologist and according to the clinical practice guidelines and standard of care, receive treatment with monoclonal antibodies against CGRP (galcanezumab, fremanezumab or eptinezumab) or else its receptor (erenumab) will be included.

Concomitant treatment:

Taking another drug with preventive purposes will be allowed as long as it is included in the national clinical practice guidelines as a preventive treatment and the drug is in a stable dose for at least 6 weeks prior to entry.

A non-probabilistic sampling will be carried out for opportunism. Patients receiving monoclonal antibody treatment in the participating centers will be included.

Intervention:

The intervention will consist of determining the time elapsed until the patients return to their pre-treatment situation once it has been suspended, at the discretion of their main neurologist or that they require a preventive treatment once again despite not having reached the pre-treatment situation. For this, the patient will be provided with an in-paper or electronic calendar in which the number of headache days, that will be completed daily. The event, also known as the month of return to the previous situation, will be defined as that month in which the number of days of pain is equal or with a difference of ± 1 day to the month prior to the start of treatment. In the event that the patient starts any preventive treatment for his migraine according to the national clinical practice guidelines, without having reached a headache frequency like the one he had before starting treatment with monoclonal antibody, it will also be classified as the event of interest.

To determine the factors that could be associated with a long-term effect, a series of variables will be assessed. Including demographic variables: sex, age, type of migraine (episodic or chronic), duration of migraine disease (in years) and duration of chronic migraine (in months). Clinical variables evaluated at the baseline level will also be analyzed: such as the number of headache days, number of migraine days, number of days of symptomatic medication, number of days of triptans, average intensity of headache on an analog verbal scale 0- 10 (0: no pain, 10: worst possible pain), MIDAS score at baseline, baseline HIT-6 score, predominance of holocranial or hemicranial, presence of periocular pain, predominant quality of pain (throbbing, pressing, stabbing, electrical) and presence of allodynia (as observed on examination or reported in the anamnesis). The number of preventive drugs previously used will be considered, understanding these as those drugs with a possible prophylactic effect for migraine, present in the local clinical practice guidelines, taken for long enough at the discretion of the responsible neurologist and at a sufficient dose or that has been suspended due to adverse effects. The dose of the monoclonal antibody used and its treatment duration in months will be evaluated.

Prior to the discontinuation of mABs, the monthly number of days with headache, migraine, symptomatic medication, triptans use, average intensity of episodes and total score of MIDAS and HIT-6 scale per month will be determined, by comparing the results obtained in the month prior to the mAbs start with the results observed in the month prior to discontinuation of treatment. It will also be described whether any adverse effect has occurred during the treatment at the discretion of the investigator.

Sample size calculation:

There is no formal sample size estimation, and all the available patients will be included.

Schedule:

The duration of the study will be of at least the next 12 months after stopping preventive treatment.

Confidentiality / Ethical aspects The study will be carried out in accordance with the precepts of the Helsinki declaration and have been approved by the Valladolid East Clinical Research Ethics Committee (PI 20-1687). All participants of the study will sign an informed consent form.

In accordance with Fundamental Law 3/2018 of December 5, Protection of Personal Data and Guarantee of Digital Rights will be respected. Be that as it may, the patient can request access, rectification, cancellation and opposition of his/her personal data. Participants will be explicitly informed that they can withdraw their participation whenever they want and reassured that they will have no disbenefit or negative effects on their future health care service from withdrawing their participation. Also, participants will be given the option to withdraw the data they have contributed with even if it is encrypted and without given any reason to request it. These will not have any economic cost for the patient. Tthe data obtained will be encoded. The password and access to it will be guarded by the researcher responsible for each center.

Possible limitations and proposed mitigations:

Observational studies are prone to biases and bias recalls, particularly when comes to filling in questionnaires. To mitigate this, participants will be trained at the beginning of study and reinforced every time is needed. Patients will have no limitations of time for completing questionaries, allowing them to complete them with the most truthful and objective information as possible; these instruments will be completed under the supervision of the research staff. Questionnaires will always be administered in the same order, beginning with the hetero-administered ones, and concluding with the self-administered ones, to avoid changes due to the fatigue effect.

Statistical analysis:

Qualitative data will be presented as frequency and percentage and in the case of quantitative data as mean and standard deviation or median and interquartile range according to the type of distribution.

To determine the principal objective, a survival analysis and determination of the Kaplan-Meier curve will be carried out to determine the probability of persistence of the effect on a monthly basis up to 12 months and its 95% confidence interval.

An analysis will be performed using the Log-Rank Test (Mantel-Cox regression) to evaluate which variables are associated with a more prolonged duration of the effect.

An alpha error of 5% will be considered and statistical compensation will be made for multiple comparisons.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with episodic or chronic migraine according to criteria of the International Classification of Headache Disorders, 3rd Edition.
2. Patients who previously received treatment with a monoclonal antibody (mABs) against CGRP or its receptor at the discretion of their usual neurologist, according to the standard of care and local guidelines.
3. Patients who experienced a positive therapeutic response to mAbs.
4. Patients that received the treatment for a minimum of 3 months.
5. Age between 18 and 65 years.
6. Participants must be capable to describe his/her clinical situation and the characteristics of his/her headache.
7. Participants must have signed the informed consent and have sufficient understanding of Spanish language.

Exclusion Criteria:

1. Presence of another type of concomitant chronic headache, defined by frequency greater than 15 days per month in the previous three months, except for medication overuse headache.
2. Patients planning to start another treatment with a possible preventive effect according to the national clinical practice guidelines within the six following weeks after their inclusion in the present study for any therapeutic indication.
3. Patients who started another treatment with a possible preventive effect according to the national clinical practice guidelines within the previous six weeks of the evaluation of the inclusion in the present study.
4. Pregnancy or breastfeeding.
5. Patients who discontinued treatment with the monoclonal antibody due to an adverse effect and not to an efficacy response.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of episodic or chronic migraine who, under the criteria of their neurologist and according to the clinical practice guidelines and standard of care, receive treatment with monoclonal antibodies against CGRP (galcanezumab, fremanezumab or eptinezumab) or else its receptor (erenumab) will be included
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Return to the baseline | Through study completion, an average of 3 months
  The needed number of months elapsed until the patient has a number of headache days per month that equals the situation at the moment of the monoclonal antibody onset, or the need of other prophylactic medication.

SECONDARY OUTCOMES:
Worsening within the first three months | Through study completion, an average of 3 months
  Determine the percentage of patients who have returned to their previous situation, or require preventive treatment once again between 15 and 90 days (3 months).
Worsening between three and six months | Through study completion, an average of 6 months
  Determine the percentage of patients who have returned to their previous situation, or require preventive treatment once again between 91 and 180 days (6 months).
Worsening between six and nine months | Through study completion, an average of 9 months
  Determine the percentage of patients who have returned to their previous situation, or require preventive treatment once again between 181 and 270 days (9 months).
Worsening between nine and twelve months | Through study completion, an average of 12 months
  Determine the percentage of patients who have returned to their previous situation, or require preventive treatment once again between 271 and 365 days (12 months).
Explore predictors of a more prolonged response | Through study completion, an average of 12 months
  Determine which demographic and clinical variables are associated with a more prolonged benefit over time.

CONTACTS AND LOCATIONS:
Overall Officials: David García Azorín, MD, PhD, Principal Investigator — Research coordinator
Locations (1):
- Hospital Clínico Universitario de Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data may be shared upon reasonable request to the principal investigator.

REFERENCES:
- [Background] Deen M, Correnti E, Kamm K, Kelderman T, Papetti L, Rubio-Beltran E, Vigneri S, Edvinsson L, Maassen Van Den Brink A; European Headache Federation School of Advanced Studies (EHF-SAS). Blocking CGRP in migraine patients - a review of pros and cons. J Headache Pain. 2017 Sep 25;18(1):96. doi: 10.1186/s10194-017-0807-1. PMID 28948500
- [Background] Edvinsson L, Haanes KA, Warfvinge K, Krause DN. CGRP as the target of new migraine therapies - successful translation from bench to clinic. Nat Rev Neurol. 2018 Jun;14(6):338-350. doi: 10.1038/s41582-018-0003-1. PMID 29691490
- [Background] Tepper S, Ashina M, Reuter U, Brandes JL, Dolezil D, Silberstein S, Winner P, Leonardi D, Mikol D, Lenz R. Safety and efficacy of erenumab for preventive treatment of chronic migraine: a randomised, double-blind, placebo-controlled phase 2 trial. Lancet Neurol. 2017 Jun;16(6):425-434. doi: 10.1016/S1474-4422(17)30083-2. Epub 2017 Apr 28. PMID 28460892
- [Background] Goadsby PJ, Reuter U, Hallstrom Y, Broessner G, Bonner JH, Zhang F, Sapra S, Picard H, Mikol DD, Lenz RA. A Controlled Trial of Erenumab for Episodic Migraine. N Engl J Med. 2017 Nov 30;377(22):2123-2132. doi: 10.1056/NEJMoa1705848. PMID 29171821
- [Background] Silberstein SD, Dodick DW, Bigal ME, Yeung PP, Goadsby PJ, Blankenbiller T, Grozinski-Wolff M, Yang R, Ma Y, Aycardi E. Fremanezumab for the Preventive Treatment of Chronic Migraine. N Engl J Med. 2017 Nov 30;377(22):2113-2122. doi: 10.1056/NEJMoa1709038. PMID 29171818
- [Background] Stauffer VL, Dodick DW, Zhang Q, Carter JN, Ailani J, Conley RR. Evaluation of Galcanezumab for the Prevention of Episodic Migraine: The EVOLVE-1 Randomized Clinical Trial. JAMA Neurol. 2018 Sep 1;75(9):1080-1088. doi: 10.1001/jamaneurol.2018.1212. PMID 29813147
- [Background] Skljarevski V, Matharu M, Millen BA, Ossipov MH, Kim BK, Yang JY. Efficacy and safety of galcanezumab for the prevention of episodic migraine: Results of the EVOLVE-2 Phase 3 randomized controlled clinical trial. Cephalalgia. 2018 Jul;38(8):1442-1454. doi: 10.1177/0333102418779543. Epub 2018 May 31. PMID 29848108
- [Background] Detke HC, Goadsby PJ, Wang S, Friedman DI, Selzler KJ, Aurora SK. Galcanezumab in chronic migraine: The randomized, double-blind, placebo-controlled REGAIN study. Neurology. 2018 Dec 11;91(24):e2211-e2221. doi: 10.1212/WNL.0000000000006640. Epub 2018 Nov 16. PMID 30446596
- [Background] Dodick DW, Ashina M, Brandes JL, Kudrow D, Lanteri-Minet M, Osipova V, Palmer K, Picard H, Mikol DD, Lenz RA. ARISE: A Phase 3 randomized trial of erenumab for episodic migraine. Cephalalgia. 2018 May;38(6):1026-1037. doi: 10.1177/0333102418759786. Epub 2018 Feb 22. PMID 29471679
- [Background] Dodick DW, Silberstein SD, Bigal ME, Yeung PP, Goadsby PJ, Blankenbiller T, Grozinski-Wolff M, Yang R, Ma Y, Aycardi E. Effect of Fremanezumab Compared With Placebo for Prevention of Episodic Migraine: A Randomized Clinical Trial. JAMA. 2018 May 15;319(19):1999-2008. doi: 10.1001/jama.2018.4853. PMID 29800211
- [Background] Ferrari MD, Diener HC, Ning X, Galic M, Cohen JM, Yang R, Mueller M, Ahn AH, Schwartz YC, Grozinski-Wolff M, Janka L, Ashina M. Fremanezumab versus placebo for migraine prevention in patients with documented failure to up to four migraine preventive medication classes (FOCUS): a randomised, double-blind, placebo-controlled, phase 3b trial. Lancet. 2019 Sep 21;394(10203):1030-1040. doi: 10.1016/S0140-6736(19)31946-4. Epub 2019 Aug 16. PMID 31427046
- [Background] Aurora SK, Winner P, Freeman MC, Spierings EL, Heiring JO, DeGryse RE, VanDenburgh AM, Nolan ME, Turkel CC. OnabotulinumtoxinA for treatment of chronic migraine: pooled analyses of the 56-week PREEMPT clinical program. Headache. 2011 Oct;51(9):1358-73. doi: 10.1111/j.1526-4610.2011.01990.x. Epub 2011 Aug 29. PMID 21883197
- [Background] Diener HC, Bussone G, Van Oene JC, Lahaye M, Schwalen S, Goadsby PJ; TOPMAT-MIG-201(TOP-CHROME) Study Group. Topiramate reduces headache days in chronic migraine: a randomized, double-blind, placebo-controlled study. Cephalalgia. 2007 Jul;27(7):814-23. doi: 10.1111/j.1468-2982.2007.01326.x. Epub 2007 Apr 18. PMID 17441971
- [Background] Pascual J, El Berdei Y, Gomez-Sanchez JC. How many migraine patients need prolonged (>1 year) preventive treatment? Experience with topiramate. J Headache Pain. 2007 Apr;8(2):90-3. doi: 10.1007/s10194-007-0351-x. Epub 2007 Jan 15. PMID 17221343
- [Background] Rapoport A, Mauskop A, Diener HC, Schwalen S, Pfeil J. Long-term migraine prevention with topiramate: open-label extension of pivotal trials. Headache. 2006 Jul-Aug;46(7):1151-60. doi: 10.1111/j.1526-4610.2006.00506.x. PMID 16866719
- [Background] Diener HC, Agosti R, Allais G, Bergmans P, Bussone G, Davies B, Ertas M, Lanteri-Minet M, Reuter U, Sanchez Del Rio M, Schoenen J, Schwalen S, van Oene J; TOPMAT-MIG-303 Investigators Group. Cessation versus continuation of 6-month migraine preventive therapy with topiramate (PROMPT): a randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2007 Dec;6(12):1054-62. doi: 10.1016/S1474-4422(07)70272-7. Epub 2007 Nov 7. PMID 17988947
- [Background] Ching J, Tinsley A, Rothrock J. Prognosis Following Discontinuation of OnabotulinumA Therapy in "Super-responding" Chronic Migraine Patients. Headache. 2019 Sep;59(8):1279-1285. doi: 10.1111/head.13630. Epub 2019 Sep 9. PMID 31498897
- [Background] Raffaelli B, Mussetto V, Israel H, Neeb L, Reuter U. Erenumab and galcanezumab in chronic migraine prevention: effects after treatment termination. J Headache Pain. 2019 Jun 3;20(1):66. doi: 10.1186/s10194-019-1018-8. PMID 31159727
- [Background] Dominguez C, Pozo-Rosich P, Torres-Ferrus M, Hernandez-Beltran N, Jurado-Cobo C, Gonzalez-Oria C, Santos S, Monzon MJ, Latorre G, Alvaro LC, Gago A, Gallego M, Medrano V, Huerta M, Garcia-Alhama J, Belvis R, Leira Y, Leira R. OnabotulinumtoxinA in chronic migraine: predictors of response. A prospective multicentre descriptive study. Eur J Neurol. 2018 Feb;25(2):411-416. doi: 10.1111/ene.13523. Epub 2017 Dec 18. PMID 29171146
- [Background] Pagola I, Esteve-Belloch P, Palma JA, Luquin MR, Riverol M, Martinez-Vila E, Irimia P. [Predictive factors of the response to treatment with onabotulinumtoxinA in refractory migraine]. Rev Neurol. 2014 Mar 16;58(6):241-6. Spanish. PMID 24610690